CLINICAL TRIAL: NCT06910072
Title: Paclitaxel Polymeric Micelles and Carboplatin in Combination With Iparomilimab and Tuvonralimab Neoadjuvant Therapy for Triple-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5182
Record Dates: First submitted 2025-02-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Triple-Negative Breast Cancer (TNBC); Neoadjuvant Therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy combined with immunotherapy (Experimental): paclitaxel polymeric micelles 300mg/m2, d1 carboplatin AUC=5, d1 iparomilimab and tuvonralimab 5mg/kg, d1 Every 3 weeks (Q3W) is a cycle, a total of 6 cycles.
  Interventions: Drug: paclitaxel polymeric micelles + carboplatin + iparomilimab and tuvonralimab

INTERVENTIONS:
Drug: paclitaxel polymeric micelles + carboplatin + iparomilimab and tuvonralimab — paclitaxel polymeric micelles 300mg/m2, d1 carboplatin AUC=5, d1 iparomilimab and tuvonralimab 5mg/kg, d1 Every 3 weeks (Q3W) is a cycle, a total of 6 cycles.

SUMMARY:
This is a prospective, single-arm, multicenter study to observe and evaluate the efficacy and safety of paclitaxel polymeric micelles and carboplatin in combination with iparomilimab and tuvonralimab in neoadjuvant therapy for triple-negative breast cancer. The main endpoint of the study is pCR, 32 patients are scheduled to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Triple-negative breast cancer
* The diameter of the primary tumor must be greater than 2cm, and the clinical stage should be II-III
* There is sufficient primary organ function
* The ECOG (PS) score is 0 or 1
* Expected survival ≥ 6 months
* The serum pregnancy test was negative. Use highly effective methods of contraception during the study period and for 180 days after the last dose of the study drug, and do not breastfeed

Exclusion Criteria:

* Bilateral breast cancer
* There is a history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS)
* A history of invasive or metastatic breast cancer
* Any malignancy diagnosed within 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or squamous cell carcinoma
* There is an immune deficiency disease
* The presence of any autoimmune disease that still requires treatment or a history of prior autoimmune disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | After surgery（within 1 month）
  Pathological complete response (pCR) rates in patients with triple-negative breast cancer

SECONDARY OUTCOMES:
Objective response rate (ORR) | During neoadjuvant therapy before surgery（within 6 months）
The rate of event-free Survival (EFS) | 2-year
The incidence of treatment-related adverse event | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No